CLINICAL TRIAL: NCT00637663
Title: Randomized, Open-Labeled Study Evaluating the Antiviral Efficacy, Safety, and Tolerability of Continuing Lamivudine Therapy or Switching to Entecavir in Subjects With Chronic Hepatitis B Who Achieved Undetectable HBV DNA
Brief Title: Continuing Lamivudine Versus Switching to Entecavir in Patients Who Achieved Undetectable Hepatitis B Virus DNA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Collaborators: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0740-67-5
Record Dates: First submitted 2008-03-04; First posted 2008-03-18 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic hepatitis B; Lamivudine; Entecavir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): entecavir 0.5 mg QD
  Interventions: Drug: Entecavir
- B (Active Comparator): lamivudine 100 mg QD
  Interventions: Drug: Lamivudine

INTERVENTIONS:
Drug: Entecavir — entecavir 0.5 mg QD
  Other Names: Baraclude 0.5mg
  Arms: A
Drug: Lamivudine — lamivudine 100 mg QD
  Other Names: Zeffix 100mg QD
  Arms: B

SUMMARY:
This is a randomized, open-labelled, prospective 96-week study comparing the antiviral efficacy and safety of switching to entecavir 0.5mg QD from lamivudine versus maintaining lamivudine 100mg QD treatment in CHB patients currently receiving lamivudine monotherapy.

DETAILED DESCRIPTION:
Entecavir has a higher potent antiviral efficacy and a lower drug resistance rate than those of Lamivudine in nucleoside-naïve CHB patients. The switch from Lamivudine to Entecavir in patients who have undetectable hepatitis B virus DNA (HBV DNA < 60 IU/mL) may lead to more prolonged viral suppression to undetectable level by PCR method, compared to patients with continuous lamivudine treatment. The results of this study will provide a rationale for switch treatment from one antiviral to another one, especially from LAM to ETV.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18-70 years of age) currently taking lamivudine monotherapy for chronic HBV infection for at least 6 months with < HBV DNA 60 IU/mL level and HBeAg positive status.

Exclusion Criteria:

* Subjects treated with other antiviral drugs (e.g. adefovir) in combination with lamivudine are not eligible for this study.
* Subjects should have ALT < 10 x ULN, and no evidence of hepatocellular carcinoma.
* Subjects should be without serological evidence of co-infection with HCV, HIV, or HDV.
* Subjects with decompensated liver disease, as well as pregnant or breast-feeding women, will not be eligible for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Percentage number of patients with HBV DNA < 60 IU/mL (Undetectable serum HBV DNA by PCR method) while on randomized therapy | at Week 96

SECONDARY OUTCOMES:
Percentage number of patients with HBV DNA < 60 IU/mL (Undetectable serum HBV DNA by PCR method) while on randomized therapy | at Week 48
Percentage number of patients who achieved ALT normalization, HBeAg loss, HBe seroconversion, HBsAg loss and HBs seroconversion | at Week 48 and 96
Cumulative discontinuation rates due to lamivudine or entecavir resistance mutations and clinical breakthrough, Safety assessment | Follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Heo, M.D. Ph.D, Study Chair — Pusan National University; Sang Hoon Ahn, M.D.Ph.D, Study Director — Yonsei Univsersity College of Medicine; Jun Yong Park, M.D, Principal Investigator — Yonsei University
Locations (2):
- South Korea (2):
  - Pusan National University School of Medicine, Busan, Busan
  - Severance Hospital, Seoul, Seoul